CLINICAL TRIAL: NCT07037290
Title: Ankle Proprioceptive Neuromuscualar Facilitation Technique Verus Foot Core Excercise in Patients With Plantar Fascitis
Brief Title: Ankle Proprioceptive Neuromuscular Facilitation Technique Versus Foot Core Exercise in Patients With Plantar Fascitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall20/1010
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Plantar Fascitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ankle proprioceptive neuromuscualar facilitation technique (Experimental)
  Interventions: Diagnostic Test: Ankle proprioceptive neuromuscualar facilitation technique
- Foot core exercises along with conventional physiotherapy (Experimental)
  Interventions: Diagnostic Test: Foot core exercises along with conventional physiotherapy

INTERVENTIONS:
Diagnostic Test: Ankle proprioceptive neuromuscualar facilitation technique — Proprioceptive Neuromuscular Facilitation (PNF) is a therapeutic technique that uses sensory input to enhance muscle function and improve flexibility. For the ankle, PNF techniques can be used to increase range of motion, improve balance and stability, and reduce pain associated with ankle injuries.
  Arms: Ankle proprioceptive neuromuscualar facilitation technique
Diagnostic Test: Foot core exercises along with conventional physiotherapy — This Group will be given foot core exercises which includes heel raise, toe curls, foot doming, toe spreading, balancing board, and tennis ball roll under foot along with conventional therapy which includes ultrasound, plantar fascia stretching and Achilles stretching.
  Arms: Foot core exercises along with conventional physiotherapy

SUMMARY:
Plantar fasciitis is a common cause of heel pain due to overuse or repetitive stress on the plantar fascia. Risk factors include abnormal foot structure, obesity, and poor footwear. Physiotherapy interventions like foot core exercises and ankle proprioceptive neuromuscular facilitation (PNF) are gaining attention for improving pain and foot function.

DETAILED DESCRIPTION:
To compare the effects of ankle PNF and foot core exercises on pain, foot posture, and function in patients with plantar fasciitis.

A randomized controlled trial will be conducted with 50 participants, divided into two groups. Group A will receive ankle PNF and Group B will receive foot core exercises, both alongside conventional physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants between 30 to 50 years of age
* Plantar fasciitis diagnosed case.
* Both males and females.
* Unilateral or bilateral involvement with acute or chronic plantar fasciitis.
* Positive windlass test.
* Patient with previous plantar fascia pain from the past 3 months.
* Patient who reported medial plantar calcaneal discomfort in initial steps after waking up.

Exclusion Criteria:

* Patients with recent history of using steroid injections or anti-inflammatory medicine use.
* Patient with any Peripheral vascular diseases
* Patients with History of fractures or gait or postural foot abnormality.
* Patients with Skin infections and wounds on the foot
* Patients with any neurological deficit involving foot
* Patients with a history of foot or ankle surgery.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
The Foot Function Index (FFI) | 6 Month
  The Foot Function Index (FFI) is a questionnaire used to assess how foot problems affect a person's daily life, specifically focusing on pain, disability, and activity limitations. It involves self-reporting scores on a scale (often 0-10 or 0-100) for various activities, with higher scores indicating greater impact.
Foot Posture Index (FPI-6) | 6 Months
  The Foot Posture Index (FPI-6) is a tool used to assess foot posture, with scores ranging from -12 (highly supinated) to +12 (highly pronated). A score between 0 and +5 is generally considered normal, while scores of +6 to +9 indicate pronation, and 10+ indicate highly pronated feet. Conversely, scores of -1 to -4 are considered supinated, and -5 to -12 are highly supinated

CONTACTS AND LOCATIONS:
Locations (1):
- Prime Care Clinic & Nazar labana, sharaqpur Sheikhupura road, near motorway interchange, Sharaqpur Sharif, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No